CLINICAL TRIAL: NCT07380490
Title: Randomised Controlled Trial Comparing the Safety and EfficAcy of the Cocoon PFO Occluder Versus Amplatzer PFO ClosurE Device for Percutaneous Closure of Patent Foramen Ovale in Patients With a History of Stroke or Transient Ischemic Attack A Non-Profit, Single-blind, Investigator Driven Trial
Brief Title: Comparing Two PFO Closure Devices in Adults With Previous Stroke or TIA
Acronym: SAFE-PFO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Giuseppe Tarantini (Industry)
Collaborators: Sahajanand Medical Technologies Limited (Industry)
Responsible Party: Sponsor-Investigator, Giuseppe Tarantini, Professor, Sahajanand Medical Technologies Limited
Organization: Sahajanand Medical Technologies Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAFE-PFO
Record Dates: First submitted 2025-11-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Patent Foramen Ovale; Stroke; Transient Ischemic Attack (TIA)
Keywords: PFO Closure; Cocoon PFO Occluder; Amplatzer PFO Occluder; Patent Foramen Ovale; Cryptogenic Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Foramen Ovale, Patent; Stroke; Ischemic Attack, Transient; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study is single-blind. Participants are masked to the device used (Cocoon vs. Amplatzer). Treating physicians and study staff involved in the procedure are not blinded due to the nature of the intervention. Participants may request unblinding at any time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cocoon PFO Occluder - experimental (Experimental): Participants undergo percutaneous closure of patent foramen ovale (PFO) using the Cocoon PFO Occluder device. The procedure is performed under standard clinical practice. Follow-up includes echocardiographic assessment of PFO closure and routine clinical evaluations. Participants are assigned to the two study arms using a 3:1 randomization scheme (Cocoon PFO Occluder : Amplatzer PFO Occluder).
  Interventions: Device: PFO Closure procedure
- Amplatzer PFO Occluder - Control (Active Comparator): Participants undergo percutaneous closure of patent foramen ovale (PFO) using the Amplatzer PFO Occluder device, considered the current standard of care. Follow-up includes echocardiographic assessment of PFO closure and routine clinical evaluations. Participants are assigned to the two study arms using a 3:1 randomization scheme (Cocoon PFO Occluder : Amplatzer PFO Occluder).
  Interventions: Device: PFO Closure procedure

INTERVENTIONS:
Device: PFO Closure procedure — Percutaneous PFO closure performed according to standard clinical practice. The procedure is scheduled within 45 days after randomization and includes initiation of dual antiplatelet therapy before the intervention. Closure is performed following the Instructions for Use (IFU) of the assigned device and is guided by intracardiac echocardiography or transesophageal echocardiography. After device implantation, patients undergo routine post-procedure assessment and are instructed to follow antiplatelet therapy consistent with European clinical practice guidelines. Endocarditis prophylaxis is recommended for six months. The procedural steps are identical for both study arms; the only difference is the device implanted (Cocoon PFO Occluder or Amplatzer PFO Occluder). Participants are assigned to the two study arms using a 3:1 randomization scheme (Cocoon PFO Occluder : Amplatzer PFO Occluder).

SUMMARY:
This study is a prospective, multicenter, randomized, controlled, single-blind, investigator-driven, non-profit clinical trial designed to compare the safety and efficacy of the Cocoon PFO Occluder with the Amplatzer PFO Occluder family in patients requiring percutaneous closure of a patent foramen ovale (PFO). Eligible participants are adults with a history of cryptogenic embolic stroke or neurologically confirmed transient ischemic attack (TIA) within the previous 12 months and a PFO suitable for transcatheter closure.

A total of up to 1260 subjects will be enrolled across multiple European centers. Participants will be randomly assigned in a 3:1 ratio to receive either the Cocoon PFO Occluder (experimental group) or an Amplatzer PFO closure device (control group). The procedure will be performed as soon as possible after randomization, preferably within 14 days and no later than 45 days.

The primary endpoint is a non-inferiority comparison of a composite outcome at 12 months, including recurrent ischemic stroke, TIA, or all-cause death. Secondary endpoints include PFO closure rate at 6 months, assessed by echocardiographic imaging, and other measures of safety, device performance, and clinical outcomes.

The study is conducted in a single-blind fashion: patients will not be informed of the device they receive unless they explicitly request this information. Any patient who chooses to be unblinded will continue to participate without affecting eligibility or follow-up, and the date of unblinding will be documented to allow appropriate sensitivity analyses.

This trial aims to provide robust comparative evidence on the clinical performance of the Cocoon PFO Occluder relative to the Amplatzer PFO Occluder to guide optimal device selection in patients with cryptogenic stroke or TIA associated with PFO.

ELIGIBILITY:
Inclusion Criteria:

* Patients with >18 years of age and <65 years of age, regardless of gender
* Patients with normal or aneurysm type PFO confirmed by imaging examination [Transthoracic Echocardiography (TTE)/ Transesophageal Echocardiography (TOE) or Intracardiac Echocardiography], and who exhibit spontaneous right-to-left shunting or right-to-left shunting during Valsalva maneuver.
* Patients with history of cryptogenic embolic stroke or transient ischemic attack in the previous 12 months [stroke is defined as acute focal neurological deficit presumed to be due to focal ischemia, and either 1) symptoms persisting 24 hours or greater, or 2) symptoms persisting less than 24 hours but associated with MR or CT findings of a new, neuroanatomically relevant, cerebral infarct. Transient Ischemic Attack is defined as acute focal neurological deficit (defined as focal motor deficit, aphasia, difficulty walking, hemisensory deficit, amaurosis fugax, blindness, or focal visual deficit) presumed due to focal ischemia, lasting between 5 minutes and 24 hours, that is not associated with MR or CT findings of a new cerebral infarct]. The diagnosis of cryptogenic embolic stroke or TIA has to be confirmed by a neurologist.
* The size of PFO must be amenable to selection of a Cocoon PFO Occluder or Amplatzer PFO closure device.
* Patients are informed of the nature of the trial and agree to all requirements for participation in the trial, signed the informed consent form, and agreed to complete the follow-up and follow-up examination

Exclusion Criteria:

* Patients who have definite causes of stroke or transient ischemic attack unrelated to the PFO
* RLS caused by other causes, such as atrial septal defect or pulmonary arteriovenous shunt
* Patients with atrial fibrillation/atrial flutter (chronic or intermittent) Intracardiac thrombus or tumor
* Patients with mitral or aortic valve stenosis or severe regurgitation
* Mitral or aortic valve vegetation or prosthesis
* Active endocarditis or other untreated infectious diseases
* Dilated cardiomyopathy, hypertrophic cardiomyopathy, restrictive cardiomyopathy
* Left ventricular ejection fraction (LVEF) <35%
* Left ventricular aneurysm or akinesis Myocardial infarction or unstable angina pectoris within 12 months
* Previous intracardiac surgery or percutaneous PFO-closure
* Atherosclerosis or arteriopathy of intra- or extracranial vessels with >50% diameter stenosis in the artery supplying the infarcted territory.
* Patients with non-embolic cryptogenic stroke (for example lacunar stroke) or with other identifiable causes of stroke, including but not limited to aortic arch plaques (protruding >4 mm into the lumen), large artery atherosclerotic disease, an established cardioembolic source, small-vessel occlusive disease, or arterial dissection
* Glomerular filtration rate < 30 ml/min/1.73 m2 or with any history of renal dialysis or renal transplantation
* Severe liver function impairment (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 times the upper limit of normal value）
* Severe pulmonary disease including pulmonary hypertension (clinical diagnosis)
* Uncontrollable hypertension or diabetes mellitus
* Contraindications to anticoagulants or antiplatelet drugs, either before or after the PFO closure procedure
* Active or planned (within 12 months) pregnancy, or lactating female patients
* Patients with hypercoagulable states
* Patients diagnosed with a neurological disease that causes progressive neurological dysfunction
* Malignant tumors or other serious diseases resulting in a life expectancy of less than 12 months
* Anatomy in which the device would interfere with intracardiac or vascular structures
* Psychiatric conditions that may interfere with medical compliance and compliance with follow-up
* Patient is currently participating in another investigational drug or device study that has not reached its primary endpoint yet
* Patient with any medical condition that would make him/her inappropriate for treatment as per the current IFU of respective devices or in the opinion of the Investigator
* Inability to obtain Informed Consent from patient or legally authorized representatives
* Stroke with poor outcome at time of enrollment (Modified Rankin score >3)
* Subjects who will not be available for follow up for the duration of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of recurrent ischemic stroke, TIA, or all-cause death at 12 months | 12 months after the procedure
  A non-inferiority comparison between the Cocoon PFO Occluder and the Amplatzer PFO Occluder in terms of a composite endpoint including:
  1. Recurrent ischemic stroke, defined as an acute focal neurological deficit presumed to result from focal ischemia, with symptoms lasting ≥24 hours, or <24 hours if accompanied by MRI or CT evidence of a new, anatomically relevant cerebral infarct.
  2. Transient ischemic attack (TIA), defined as an acute focal neurological deficit (e.g., focal motor deficit, aphasia, gait disturbance, hemisensory deficit, amaurosis fugax, blindness, or focal visual deficit) presumed due to focal ischemia, lasting between 5 minutes and 24 hours, and not associated with MRI or CT evidence of a new infarct. Clinical evaluation by a neurologist is required.
  3. All-cause mortality.

SECONDARY OUTCOMES:
PFO Closure Rate | 6 months
  Complete closure is defined as right-to-left shunt (RLS) grade 0. Effective closure is defined as RLS grade 0 or 1 on imaging (TTE as default, TOE when clinically indicated)
Composite of Recurrent Ischemic Stroke, TIA, or Death | 30 days and 6 months
  Composite endpoint including recurrent ischemic stroke, TIA (neurologist-confirmed), or all-cause mortality.
Neurological Death | 30 days, 6 months, 12 months
  Death attributable to neurological causes.
Cardiovascular Death | 30 days, 6 months, 12 months
  Death attributable to cardiovascular causes.
Recurrent Symptomatic Non-Fatal Stroke | 30 days, 6 months, 12 months
  TIA defined according to the same criteria as the primary endpoint and confirmed by a neurologist
Serious Adverse Events (SAE) | 30 days, 6 months, 12 months
  Incidence of any serious adverse event as defined by standard reporting criteria.
Device- or Procedure-Related Serious Adverse Events | 30 days, 6 months, 12 months
  SAE related to the device or procedure, including but not limited to: death, systemic embolism, device embolization or malposition, device thrombosis, cardiac injury/perforation, pericardial tamponade/effusion, endocarditis, atrial fibrillation, and severe vascular access complications
Clinically Significant New Atrial Arrhythmia | 30 days, 6 months, 12 months
  New atrial arrhythmia (including AF) confirmed by ECG, Holter, or approved monitoring device. AF defined per international guidelines (≥30-second episode with absence of P waves and irregular RR intervals).
Device Success | Immediately after the procedure
  Successful delivery, deployment at intended site, and retrieval of the delivery system.
Procedural Success | At hospital discharge
  Device success without device- or procedure-related SAE prior to discharge
Change in Monthly Migraine Days | Months 9-12 vs. baseline (3 months before implantation)
  Change in monthly migraine days in patients with a neurologist-confirmed diagnosis of migraine.
Quality of Life (SF-36 Score) | 6 months, 12 months
  Assessment of quality of life using the SF-36 questionnaire.
Systemic Embolism | 30 days, 6 months, 12 months
  Incidence of systemic embolic events confirmed clinically or by imaging
Possible/Probable Device-Related Allergy | 12 months
  Device-related allergic reactions adjudicated by the Clinical Events Committee (CEC)
Echocardiographic Markers of Device Endothelialization | At 6 months (±1 month) post-procedure At 12 months (±2 months) post-procedure Additional TOE as clinically indicated through study completion (up to 12 months)
  Evaluation of endothelialization using surrogate TOE markers: device surface echogenicity, peri-device flow, presence of thrombus/mass, visible disc surface area, and bubble contrast washout. Data will be summarized as the proportion of participants meeting criteria for complete endothelialization at each follow-up time point.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Testa L, Popolo Rubbio A, Squillace M, Albano F, Cesario V, Casenghi M, Tarantini G, Pagnotta P, Ielasi A, Popusoi G, Paloscia L, Durante A, Maffeo D, Meucci F, Valentini G, Ussia GP, Cioffi P, Cortese B, Sangiorgi G, Contegiacomo G, Bedogni F. Patent foramen ovale occlusion with the Cocoon PFO Occluder. The PROS-IT collaborative project. Front Cardiovasc Med. 2023 Jan 11;9:1064026. doi: 10.3389/fcvm.2022.1064026. eCollection 2022. PMID 36712245
- [Background] Turc G, Calvet D, Guerin P, Sroussi M, Chatellier G, Mas JL; CLOSE Investigators. Closure, Anticoagulation, or Antiplatelet Therapy for Cryptogenic Stroke With Patent Foramen Ovale: Systematic Review of Randomized Trials, Sequential Meta-Analysis, and New Insights From the CLOSE Study. J Am Heart Assoc. 2018 Jun 17;7(12):e008356. doi: 10.1161/JAHA.117.008356. PMID 29910193
- [Background] Lee PH, Song JK, Kim JS, Heo R, Lee S, Kim DH, Song JM, Kang DH, Kwon SU, Kang DW, Lee D, Kwon HS, Yun SC, Sun BJ, Park JH, Lee JH, Jeong HS, Song HJ, Kim J, Park SJ. Cryptogenic Stroke and High-Risk Patent Foramen Ovale: The DEFENSE-PFO Trial. J Am Coll Cardiol. 2018 May 22;71(20):2335-2342. doi: 10.1016/j.jacc.2018.02.046. Epub 2018 Mar 12. PMID 29544871
- [Background] Mas JL, Derumeaux G, Guillon B, Massardier E, Hosseini H, Mechtouff L, Arquizan C, Bejot Y, Vuillier F, Detante O, Guidoux C, Canaple S, Vaduva C, Dequatre-Ponchelle N, Sibon I, Garnier P, Ferrier A, Timsit S, Robinet-Borgomano E, Sablot D, Lacour JC, Zuber M, Favrole P, Pinel JF, Apoil M, Reiner P, Lefebvre C, Guerin P, Piot C, Rossi R, Dubois-Rande JL, Eicher JC, Meneveau N, Lusson JR, Bertrand B, Schleich JM, Godart F, Thambo JB, Leborgne L, Michel P, Pierard L, Turc G, Barthelet M, Charles-Nelson A, Weimar C, Moulin T, Juliard JM, Chatellier G; CLOSE Investigators. Patent Foramen Ovale Closure or Anticoagulation vs. Antiplatelets after Stroke. N Engl J Med. 2017 Sep 14;377(11):1011-1021. doi: 10.1056/NEJMoa1705915. PMID 28902593
- [Background] Carroll JD, Saver JL, Thaler DE, Smalling RW, Berry S, MacDonald LA, Marks DS, Tirschwell DL; RESPECT Investigators. Closure of patent foramen ovale versus medical therapy after cryptogenic stroke. N Engl J Med. 2013 Mar 21;368(12):1092-100. doi: 10.1056/NEJMoa1301440. PMID 23514286
- [Background] Meier B, Kalesan B, Mattle HP, Khattab AA, Hildick-Smith D, Dudek D, Andersen G, Ibrahim R, Schuler G, Walton AS, Wahl A, Windecker S, Juni P; PC Trial Investigators. Percutaneous closure of patent foramen ovale in cryptogenic embolism. N Engl J Med. 2013 Mar 21;368(12):1083-91. doi: 10.1056/NEJMoa1211716. PMID 23514285
- [Background] Furlan AJ, Reisman M, Massaro J, Mauri L, Adams H, Albers GW, Felberg R, Herrmann H, Kar S, Landzberg M, Raizner A, Wechsler L; CLOSURE I Investigators. Closure or medical therapy for cryptogenic stroke with patent foramen ovale. N Engl J Med. 2012 Mar 15;366(11):991-9. doi: 10.1056/NEJMoa1009639. PMID 22417252
- [Background] Pristipino C, Sievert H, D'Ascenzo F, Mas JL, Meier B, Scacciatella P, Hildick-Smith D, Gaita F, Toni D, Kyrle P, Thomson J, Derumeaux G, Onorato E, Sibbing D, Germonpre P, Berti S, Chessa M, Bedogni F, Dudek D, Hornung M, Zamorano J; European Association of Percutaneous Cardiovascular Interventions (EAPCI); European Stroke Organisation (ESO); European Heart Rhythm Association (EHRA); European Association for Cardiovascular Imaging (EACVI); Association for European Paediatric and Congenital Cardiology (AEPC); ESC Working group on GUCH; ESC Working group on Thrombosis; European Haematological Society (EHA). European position paper on the management of patients with patent foramen ovale. General approach and left circulation thromboembolism. EuroIntervention. 2019 Jan 20;14(13):1389-1402. doi: 10.4244/EIJ-D-18-00622. No abstract available. PMID 30141306